CLINICAL TRIAL: NCT00876187
Title: A RANDOMIZED, DOUBLE-BLIND, MULTI-DOSE, ACTIVE- AND PLACEBO-CONTROLLED, MULTI-CENTER, PARALLEL GROUP STUDY OF THE ANALGESIC EFFECTS OF TANEZUMAB IN ADULT PATIENTS WITH CHRONIC LOW BACK PAIN
Brief Title: A Study of Tanezumab in Adults With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4091012; CLBP-IV PH2B (Other: Alias Study Number)
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain
Keywords: randomized controlled trial; monoclonal antibody; nerve growth factor; naproxen
MeSH Terms: conditions — Low Back Pain; Hereditary Sensory and Autonomic Neuropathies | interventions — tanezumab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Tanezumab 20 mg IV (Experimental)
  Interventions: Biological: Tanezumab 20 mg IV; Drug: Placebo for naproxen
- Tanezumab 10 mg IV (Experimental)
  Interventions: Biological: Tanezumab 10 mg IV; Drug: Placebo for naproxen
- Tanezumab 5 mg IV (Experimental)
  Interventions: Biological: Tanezumab 5 mg IV; Drug: Placebo for naproxen
- Naproxen (Active Comparator)
  Interventions: Biological: Placebo for tanezumab; Drug: Naproxen
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo for tanezumab; Drug: Placebo for naproxen

INTERVENTIONS:
Biological: Tanezumab 20 mg IV — 2 IV administrations of tanezumab 20 mg at an 8 week interval
  Arms: Tanezumab 20 mg IV
Drug: Placebo for naproxen — Oral placebo for naproxen twice a day for 16 weeks
  Arms: Tanezumab 20 mg IV
Biological: Tanezumab 10 mg IV — 2 IV administrations of tanezumab 10 mg at an 8 week interval
  Arms: Tanezumab 10 mg IV
Drug: Placebo for naproxen — Oral placebo for naproxen twice a day for 16 weeks
  Arms: Tanezumab 10 mg IV
Biological: Tanezumab 5 mg IV — 2 IV administrations of tanezumab 5 mg at an 8 week interval
  Arms: Tanezumab 5 mg IV
Drug: Placebo for naproxen — Oral placebo for naproxen twice a day for 16 weeks
  Arms: Tanezumab 5 mg IV
Biological: Placebo for tanezumab — 2 IV administrations of placebo for tanezumab at an 8 week interval
  Arms: Naproxen
Drug: Naproxen — Oral naproxen 500 mg twice a day for 16 weeks
  Arms: Naproxen
Biological: Placebo for tanezumab — 2 IV administrations of placebo for tanezumab at an 8 week interval
  Arms: Placebo
Drug: Placebo for naproxen — Oral placebo for naproxen twice a day for 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of multiple doses of tanezumab administered every 8 weeks in treating chronic low back pain. Tanezumab is a monoclonal antibody directed against human nerve growth factor.

ELIGIBILITY:
Inclusion Criteria:

* Present with duration of low back pain of ≥3 months requiring regular use of analgesic medication (>4 days per week for the past month). Analgesic medication may consist of NSAIDs, selective COX-2 inhibitors, immediate release opioids, or combinations, with certain protocol-defined limitations.
* Primary location of low back pain must be between the 12th thoracic vertebra and the lower gluteal folds, with or without radiation into the posterior thigh
* Must meet criteria for pain severity and global assessment of low back pain at Screening and Baseline visits
* Female patients of child-bearing potential (and male patients with female partners who are of child-bearing potential) must use 2 methods of contraception throughout the study
* Patients must be willing to discontinue all pain medications for chronic low back pain except rescue medication and not use prohibited pain medications throughout the duration of the study

Exclusion Criteria:

* History of lumbosacral radiculopathy within the past 2 years.
* Back pain due to visceral disorder (eg, endometriosis).
* Back pain due to major trauma or osteoporotic compression fracture in the past 6 months.
* History of rheumatoid arthritis, seronegative spondyloarthropathy, Paget's disease of spine, pelvis or femur; fibromyalgia; tumors or infections of the spinal cord.
* Surgical intervention during the past 6 months for the treatment of low back pain or plans for surgical intervention during the course of the study.
* Current or pending worker's compensation, litigation, disability, or any other monetary settlement regarding his/her CLBP or any other pain condition, or any closed claim within the past 5 years.
* Use of any analgesic or muscle relaxant within 48 hours prior to the five days before Baseline
* Patients receiving only acetaminophen, gabapentin or pregabalin to manage their chronic low back pain.
* Patients taking >325 mg/day of aspirin.
* Use of any antidepressants with the exception of stable treatment with selective serotonin reuptake inhibitors (SSRIs).
* Use of any sedatives/hypnotics, anxiolytics, tranquilizers, or benzodiazepines unless daily dose has been stable and will remain unchanged throughout the study period.
* Systemic corticosteroid therapy within 30 days (inhaled and topical corticosteroids are permitted).
* Local or epidural injection of corticosteroids, as well as injections of corticosteroids in the back within 3 months.
* Botulinum toxin (Botox®) injection for chronic low back pain within 4 months.
* Requirement for new, concomitant physiotherapy including, but not limited to, transdermal electroneural stimulation (TENS), massage or spinal manipulation for the duration of the study period.
* Active or suspected esophageal, gastric, pyloric channel, or duodenal ulceration within 3 months, or any history of gastrointestinal bleeding.
* Current use of lithium or anticoagulant agents.
* Known hypersensitivity or intolerance to NSAIDs; history of asthma, urticaria, or allergic type reactions after taking aspirin or NSAIDs.
* Inflammatory bowel disease, a chronic or acute renal or hepatic disorder, a significant coagulation defect, or other condition that might preclude the use of an NSAID.
* History of intolerance to acetaminophen or paracetamol or any of its excipients.
* History of known alcohol, analgesic or narcotic abuse within 2 years.
* Presence of drugs of abuse (including prescription medications without a valid prescription), other illegal drugs or marijuana in the urine toxicology screen obtained at Screening.
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein.
* Use of biologics other than study medication, including any live vaccines, within 3 months, or use during the study (intranasal Flumist® vaccine is an exception).
* Signs and symptoms of clinically significant cardiac disease.
* Diagnosis of a transient ischemic attack within the 6 months, or residual deficits from stroke that would preclude completion of required study activities.
* History of cancer within 5 years.
* Use of any investigational medication within 30 days (3 months for investigational biologics).
* Expected to undergo a therapeutic procedure or to use any analgesic other than those specified in the protocol throughout the study period.
* Previous exposure to exogenous NGF or to an anti NGF antibody.
* Screening laboratory results and blood pressure within specified limits.
* Positive Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) tests at screening.
* History, diagnosis, or signs and symptoms of clinically significant neurological disease.
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder.
* Hospital admission for depression or suicide attempt within 5 years or active, severe major depression at Screening.
* Likelihood of being non compliant with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1359 (Actual)
Dates: Start 2009-06-15 (Actual); Primary Completion 2010-06-16 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (133):
- United States (133):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Simon Williamson Clinic, PC, Birmingham, Alabama
  - Simon-Williamson Clinic, PC, Hueytown, Alabama
  - Saadat Ansari, MD office, Huntsville, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Radiant Research - Phoenix Southeast, Chandler, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Radiant Research, Inc.: Scottsdale, AZ, Scottsdale, Arizona
  - Premiere Phamaceutical Research, LLC, Tempe, Arizona
  - Clinical Research Advantage, Inc./Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - Alta Clinical Research, LLC, Tucson, Arizona
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - Providence Clinical Research, Burbank, California
  - Valley Research, Fresno, California
  - Collaborative Neuroscience Network, Inc, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Samaritan Center for Medical Research Medical Group, Los Gatos, California
  - North County Clinical Research (NCCR), Oceanside, California
  - Advances in Medicine, Rancho Mirage, California
  - Quality Control Research, Inc, Roseville, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Wetlin Research Associates, Inc, San Diego, California
  - Inland Rheumatology & Osteoporosis Medical Group, Inc., Upland, California
  - Elite Clinical Trials, Wildomar, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Clinicos, LLC, Colorado Springs, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - Southeast Clinical Research, Chiefland, Florida
  - Doctors Medical Center of Walton County, DeFuniak Springs, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - CRIA Research, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Compass Research, LLC, Orlando, Florida
  - University Clinical Research Incorporated, Pembroke Pines, Florida
  - Advent Clinical Research Center, Pinellas Park, Florida
  - Arthntis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Dale G. Bramlet, MD, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Center for Prospective Outcome Studies, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Drug Studies America, Marietta, Georgia
  - Selah Medical Center, PA, Boise, Idaho
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Vince and Associates Clinical Research, Overiand Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Cotton-O'Neil Clinical Research, Topeka, Kansas
  - Central Kentucky Research Association, Inc., Lexington, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Peter A. Holt, MD, Baltimore, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - PCM Medical Services, Lansing, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Clinical Research Center of Jackson, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Clinvest/ A Division of Banyan Group, Inc., Springfield, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - CRI Worldwide, Willingboro, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Medex Healthcare Research, Inc., New York, New York
  - Medex Healthcare Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Pharmquest, Greensboro, North Carolina
  - Northstate Clinical Research, PLLC, Lenoir, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Sterling Research, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Christine Codding, MD, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - McBride Clinic, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Columbia Arthritis Center, P.A., Columbia, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Radiant Research, Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - SCRI Research Center, Germantown, Tennessee
  - Wolf River Medical Group, LLC, Germantown, Tennessee
  - Advanced Therapeutics, Inc., Johnson City, Tennessee
  - Johnson City Internal Medicine, Johnson City, Tennessee
  - Capitol Medical Clinic, Austin, Texas
  - Walter F. Chase, MD, PA, Austin, Texas
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - DiscoveResearch, Incorporated, Bryan, Texas
  - Trinity Hypertension & Metabolic Research Institute Punzi Medical Center, Carrollton, Texas
  - KRK Medical Research, Dallas, Texas
  - Advances In Health, Inc., Houston, Texas
  - Centex Research, Inc., Houston, Texas
  - Centex Research, Houston, Texas
  - Centex Research, Nassau Bay, Texas
  - Office of Theresia Lee, MD, San Antonio, Texas
  - Paragon Research Center, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research, Incorporated, Richmond, Virginia
  - Advanced Pain Management, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- [Derived] Kivitz AJ, Gimbel JS, Bramson C, Nemeth MA, Keller DS, Brown MT, West CR, Verburg KM. Efficacy and safety of tanezumab versus naproxen in the treatment of chronic low back pain. Pain. 2013 Jul;154(7):1009-21. doi: 10.1016/j.pain.2013.03.006. Epub 2013 Mar 14. PMID 23628600
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091012&StudyName=A%20Study%20of%20Tanezumab%20in%20Adults%20with%20Chronic%20Low%20Back%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent for a 5-day initial pain assessment period prior to randomization.
Pre-assignment Details: Participants who discontinued due to lack of efficacy or completed the treatment in this study were eligible to enroll in safety extension study A4091039 (NCT00924664).
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over a 5-minute period at Day 1 and Week 8 along with placebo matched to naproxen tablet orally twice daily up to Week 16.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 milligram (mg) intravenous infusion over a 5-minute period at Day 1 and Week 8 along with placebo matched to naproxen tablet orally twice daily up to Week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119)10 mg intravenous infusion over a 5-minute period at Day 1 and Week 8 along with placebo matched to naproxen tablet orally twice daily up to Week 16.
- Tanezumab 20 mg: Tanezumab (RN624 or PF-04383119) 20 mg intravenous infusion over a 5-minute period at Day 1 and Week 8 along with placebo matched to naproxen tablet orally twice daily up to Week 16.
- Naproxen 500 mg: Naproxen 500 mg tablet orally twice daily up to Week 16 along with placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over a 5-minute period at Day 1 and Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Started | 233 | 233 | 298 | 297 | 298
Treated | 230 | 232 | 295 | 295 | 295
Completed Treatment | 128 (Participants who completed treatment at Week 16 visit.) | 146 (Participants who completed treatment at Week 16 visit.) | 193 (Participants who completed treatment at Week 16 visit.) | 188 (Participants who completed treatment at Week 16 visit.) | 185 (Participants who completed treatment at Week 16 visit.)
Completed | 23 | 18 | 19 | 22 | 27
Not Completed | 210 | 215 | 279 | 275 | 271
Not completed — Adverse Event | 14 | 12 | 19 | 29 | 10
Not completed — Lack of Efficacy | 59 | 34 | 45 | 34 | 59
Not completed — Lost to Follow-up | 9 | 10 | 8 | 8 | 11
Not completed — Protocol Violation | 6 | 7 | 7 | 6 | 3
Not completed — Withdrawal by Subject | 16 | 26 | 32 | 38 | 37
Not completed — Entered extension study | 101 | 120 | 156 | 151 | 144
Not completed — Randomized but not treated | 3 | 1 | 3 | 2 | 3
Not completed — Other | 2 | 5 | 9 | 7 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who received at least 1 dose of intravenous study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg | Total
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295 | 1347
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.2) | 51.5 (14.2) | 52.0 (13.9) | 51.2 (12.9) | 52.6 (13.2) | 51.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 115 | 157 | 165 | 152 | 714
  Male | 105 | 117 | 138 | 130 | 143 | 633

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 16: Baseline Observation Carried Forward (BOCF)
Description: Daily average back pain was assessed on an 11-point numeric rating scale (NRS) captured through an interactive voice response system (IVRS). The participant described the chronic low back pain (CLBP) during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain). Baseline value was calculated as mean of the scores over 5 days prior to randomization (initial pain assessment period). Post-baseline value was calculated as mean of the scores over the 7-day period prior to and including the post-baseline visit. Overall possible score range for daily average LBPI at specified visit was 0= no pain to 10= worst possible pain, where higher scores indicated higher pain intensity.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication. BOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
units on a scale
  Baseline | 6.71 (1.37) | 6.62 (1.36) | 6.57 (1.39) | 6.74 (1.48) | 6.77 (1.38)
  Change at Week 16 | -1.25 (2.01) | -1.55 (2.07) | -2.02 (2.40) | -2.19 (2.52) | -1.70 (2.28)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg; Treatment difference and 95 percent (%) confidence interval (CI) was based on least squares (LS) mean. Analysis of Covariance (ANCOVA) was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.113, ANCOVA; Least Squares (LS) Mean Difference = -0.33, 95% CI 2-sided [-0.74 to 0.08], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg; Treatment difference and 95% CI was based on LS mean. ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.80, 95% CI 2-sided [-1.19 to -0.42], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.31 to -0.54], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs Naproxen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.688, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.31 to 0.47], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Tanezumab 10 mg vs Naproxen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.035, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.76 to -0.03], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Tanezumab 20 mg vs Naproxen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.88 to -0.15], Standard Error of Mean 0.19

2. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: RMDQ: back-specific, participant administered questionnaire that assesses how well participants with low back pain were able to function with regard to daily activities. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement if it describes his/her functional ability on the day of assessment. The number of statements marked are added up by the clinician. Total RMDQ score is calculated as the sum of number of statements marked. Total possible RMDQ score: 0 (best functioning) to 24 (worst functioning), with higher scores indicated greater disability.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication. BOCF method was used to impute missing values. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 228 | 232 | 295 | 295 | 295
units on a scale
  Baseline | 12.79 (4.74) | 12.24 (4.92) | 12.98 (5.11) | 13.00 (4.97) | 12.86 (4.93)
  Change at Week 2 | -1.68 (3.74) | -2.47 (4.61) | -2.59 (4.41) | -2.39 (4.61) | -2.28 (4.19)
  Change at Week 4 | -1.85 (4.04) | -2.81 (4.52) | -3.45 (4.90) | -3.35 (4.87) | -2.39 (4.24)
  Change at Week 8 | -1.86 (4.13) | -2.62 (4.43) | -2.93 (4.75) | -3.47 (5.17) | -2.27 (4.12)
  Change at Week 12 | -1.91 (4.13) | -2.23 (3.82) | -3.16 (4.97) | -3.26 (4.81) | -2.44 (4.12)
  Change at Week 16 | -1.76 (4.15) | -2.27 (4.07) | -3.20 (5.07) | -2.82 (4.65) | -2.08 (3.85)

3. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Low Back Pain Score at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all ways your low back pain affects you, how are you doing today?" Participants rated their condition using scale assessing symptoms and limitations to carry out normal daily activities. Score range:1 to 5. 1: Very Good (No symptoms and limitations); 2: Good (Mild symptoms and no limitations); 3: Fair (Moderate symptoms and some limitations); 4: Poor (Severe symptoms and inability to carry out most activities); 5: Very Poor (Very severe, intolerable symptoms and inability to carry all activities).
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 229 | 232 | 295 | 294 | 295
units on a scale
  Baseline | 3.41 (0.58) | 3.41 (0.60) | 3.33 (0.56) | 3.36 (0.56) | 3.35 (0.56)
  Change at Week 2 | -0.55 (0.80) | -0.62 (0.91) | -0.66 (0.89) | -0.62 (1.00) | -0.59 (0.84)
  Change at Week 4 | -0.53 (0.88) | -0.78 (0.89) | -0.77 (0.90) | -0.84 (0.95) | -0.67 (0.90)
  Change at Week 8 | -0.52 (0.84) | -0.66 (0.93) | -0.71 (0.92) | -0.78 (0.93) | -0.54 (0.87)
  Change at Week 12 | -0.48 (0.82) | -0.69 (0.91) | -0.73 (0.90) | -0.74 (0.98) | -0.59 (0.86)
  Change at Week 16 | -0.42 (0.78) | -0.59 (0.96) | -0.63 (0.91) | -0.67 (0.93) | -0.49 (0.86)

4. Secondary Outcome: Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: Daily average back pain was assessed on an 11-point numeric rating scale (NRS) captured through an interactive voice response system (IVRS). The participant described the chronic low back pain (CLBP) during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain). Baseline value was calculated as mean of the scores over 5 days prior to randomization (initial pain assessment period). Post-baseline value was calculated as mean of the scores over the 7-day period prior to and including the post-baseline visit.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
units on scale
  Change at Week 2 | -1.29 (1.84) | -1.48 (1.79) | -1.83 (1.89) | -1.68 (2.19) | -1.85 (1.98)
  Change at Week 4 | -1.50 (1.95) | -1.94 (2.00) | -2.47 (2.22) | -2.44 (2.33) | -2.05 (2.05)
  Change at Week 8 | -1.40 (2.05) | -1.82 (1.99) | -2.23 (2.25) | -2.32 (2.40) | -1.82 (2.05)
  Change at Week 12 | -1.49 (2.14) | -1.92 (2.17) | -2.27 (2.47) | -2.37 (2.56) | -1.93 (2.29)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 2: Treatment difference and 95% CI was based on LS mean. ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.221, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.57 to 0.13], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.90 to -0.24], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.027, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.70 to -0.04], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.082, ANCOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.04 to 0.62], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Tanezumab 10 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.703, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.37 to 0.25], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Tanezumab 20 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.379, ANCOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.17 to 0.45], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 4: Treatment difference and 95% CI was based on LS mean. ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.87 to -0.11], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.03, 95% CI 2-sided [-1.39 to -0.67], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.94, 95% CI 2-sided [-1.31 to -0.58], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.862, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.33 to 0.39], Standard Error of Mean 0.18
Statistical Analysis 11: Comparison: Tanezumab 10 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.85 to -0.17], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Tanezumab 20 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.014, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.76 to -0.09], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 8: Treatment difference and 95% CI was based on LS mean. ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.019, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.86 to -0.08], Standard Error of Mean 0.20
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.25 to -0.51], Standard Error of Mean 0.19
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.29 to -0.56], Standard Error of Mean 0.19
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.668, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.45 to 0.29], Standard Error of Mean 0.19
Statistical Analysis 17: Comparison: Tanezumab 10 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.84 to -0.15], Standard Error of Mean 0.18
Statistical Analysis 18: Comparison: Tanezumab 20 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-0.88 to -0.19], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 12: Treatment difference and 95% CI was based on LS mean. ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.89 to -0.04], Standard Error of Mean 0.22
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.21 to -0.41], Standard Error of Mean 0.20
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.28 to -0.48], Standard Error of Mean 0.20
Statistical Analysis 22: Comparison: Tanezumab 5 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.773, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.46 to 0.34], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Tanezumab 10 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.035, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.78 to -0.03], Standard Error of Mean 0.19
Statistical Analysis 24: Comparison: Tanezumab 20 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.014, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.85 to -0.10], Standard Error of Mean 0.19

5. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline at Week 16 in Daily Average Low Back Pain Intensity (LBPI) Score : Baseline Observation Carried Forward (BOCF)
Description: Daily average back pain was assessed on an 11-point numeric rating scale (NRS) captured through an interactive voice response system (IVRS). The participant described the chronic low back pain (CLBP) during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain). Baseline value was calculated as mean of the scores over 5 days prior to randomization (initial pain assessment period). Post-baseline value was calculated as mean of the scores over the 7-day period prior to and including the post-baseline visit. Participants with specified reduction (as percent) from baseline at Week 16 are reported.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
Participants
  Greater than (>) 0% | 103 | 121 | 171 | 174 | 160
  Greater than or equal to (>=)10% | 90 | 111 | 159 | 162 | 146
  >= 20% | 78 | 99 | 136 | 145 | 128
  >= 30% | 62 | 83 | 123 | 137 | 111
  >= 40% | 53 | 64 | 112 | 120 | 92
  >= 50% | 39 | 59 | 94 | 104 | 78
  >= 60% | 31 | 42 | 78 | 80 | 60
  >= 70% | 22 | 29 | 62 | 54 | 37
  >= 80% | 12 | 24 | 45 | 40 | 26
  >= 90% | 8 | 12 | 30 | 26 | 16
  = 100% | 5 | 9 | 20 | 16 | 9

6. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%) and 50% Reduction From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 4
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
percentage of participants
  Week 2: >=30% reduction | 27.4 | 32.8 | 42.4 | 41.0 | 39.0
  Week 2: >=50% reduction | 11.3 | 20.7 | 19.3 | 22.0 | 24.4
  Week 4: >=30% reduction | 33.9 | 43.5 | 54.2 | 52.5 | 42.0
  Week 4: >=50% reduction | 16.5 | 28.9 | 35.6 | 35.9 | 25.8
  Week 8: >=30% reduction | 32.2 | 43.1 | 48.1 | 50.8 | 39.7
  Week 8: >=50% reduction | 18.7 | 25.4 | 32.5 | 35.3 | 22.7
  Week 12: >=30% reduction | 31.3 | 42.7 | 48.1 | 50.5 | 42.7
  Week 12: >=50% reduction | 22.2 | 31.0 | 36.3 | 40.0 | 30.8
  Week 16: >=30% reduction | 27.0 | 35.8 | 41.7 | 46.4 | 37.6
  Week 16: >=50% reduction | 17.0 | 25.4 | 31.9 | 35.3 | 26.4

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Score for Worst and Average Pain at Week 2, 4, 8, 12, 16: Baseline Observation Carried Forward (BOCF)
Description: BPI-sf: self-report questionnaire rated on an 11-point scale, consists of 5 questions to assess severity and impact of pain on daily functions. Question 1-4 (Q1-Q4) measure severity of pain (worst, least, average, right now), each question ranging between 0 (no pain) to 10 (pain as bad as you can imagine). Question 5 (Q5) consists of 7 items which measure level of interference of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life), each item ranging from 0 (does not interfere) to 10 (completely interferes). Results are reported for worst and average pain, each with a score range: 0 (no pain) and 10 (pain as bad as you can imagine), higher scores indicated worse pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 228 | 232 | 295 | 295 | 294
units on a scale
  Baseline: Worst Pain | 7.27 (1.51) | 7.10 (1.53) | 7.04 (1.49) | 7.36 (1.59) | 7.28 (1.51)
  Baseline: Average Pain | 6.22 (1.44) | 6.25 (1.51) | 6.08 (1.52) | 6.35 (1.45) | 6.27 (1.41)
  Change at Week 2: Worst Pain | -1.63 (2.33) | -1.76 (2.14) | -2.19 (2.41) | -2.08 (2.60) | -1.97 (2.38)
  Change at Week 2: Average Pain | -1.16 (1.93) | -1.43 (1.91) | -1.69 (2.11) | -1.65 (2.34) | -1.57 (2.07)
  Change at Week 4: Worst Pain | -1.63 (2.38) | -2.21 (2.28) | -2.57 (2.50) | -2.88 (2.64) | -2.16 (2.50)
  Change at Week 4: Average Pain | -1.19 (1.95) | -1.88 (1.91) | -2.09 (2.18) | -2.32 (2.34) | -1.77 (2.10)
  Change at Week 8: Worst Pain | -1.54 (2.33) | -1.94 (2.30) | -2.35 (2.45) | -2.55 (2.70) | -1.98 (2.31)
  Change at Week 8: Average Pain | -1.19 (1.93) | -1.78 (1.99) | -1.98 (2.18) | -2.18 (2.42) | -1.61 (1.97)
  Change at Week 12: Worst Pain | -1.63 (2.43) | -1.99 (2.41) | -2.53 (2.73) | -2.70 (2.84) | -2.13 (2.55)
  Change at Week 12: Average Pain | -1.32 (2.12) | -1.75 (2.11) | -2.13 (2.35) | -2.26 (2.54) | -1.73 (2.13)
  Change at Week 16: Worst Pain | -1.55 (2.35) | -1.75 (2.34) | -2.20 (2.66) | -2.36 (2.78) | -1.94 (2.49)
  Change at Week 16: Average Pain | -1.20 (1.95) | -1.58 (2.14) | -1.89 (2.37) | -2.03 (2.47) | -1.66 (2.19)

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Score for Pain Interference Index, Pain Interference Score for General Activity, Walking Ability, Sleep and Normal Work at Week 2, 4, 8, 12 and 16: BOCF
Description: BPI-sf: self-report questionnaire rated on an 11-point scale, consists of 5 questions to assess severity and impact of pain on daily functions. Question 1-4 (Q1-Q4) measure severity of pain (worst, least, average, right now), each question ranging between 0 (no pain) to 10 (pain as bad as you can imagine). Question 5 (Q5) consists of 7 items which measure pain interference (PI) on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life), each item ranging from 0 (does not interfere) to 10 (completely interferes); higher score = greater impairment. The 7 items in Q5 averaged to obtain pain interference index (function composite score), range: 0 (no interference) to 10 (complete interference); higher score = greater impairment.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: ITT analysis set. BOCF method was used to impute missing values. Here, "Overall number of participants analyzed" = participants who were evaluable for this outcome measure and 'Number Analyzed' = participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 228 | 231 | 295 | 295 | 295
units on a scale
  Change at Week 2: Pain Interference Index | -1.33 (2.20) | -1.59 (2.14) | -1.97 (2.33) | -1.81 (2.63) | -1.75 (2.46)
  Change at Week 4: Pain Interference Index | -1.48 (2.19) | -1.99 (2.12) | -2.40 (2.31) | -2.63 (2.44) | -2.01 (2.34)
  Change at Week 12: Pain Interference Index | -1.38 (2.19) | -1.62 (2.21) | -2.21 (2.47) | -2.38 (2.60) | -1.81 (2.39)
  Change at Week 16: Pain Interference Index | -1.32 (2.01) | -1.52 (2.19) | -2.02 (2.48) | -2.17 (2.44) | -1.59 (2.28)
  Change at Week 8: Pain Interference Index | -1.33 (2.20) | -1.65 (2.16) | -2.15 (2.34) | -2.37 (2.45) | -1.71 (2.22)
  Change at Week 2: General Activity: number analyzed (Participants) | 228 | 231 | 295 | 295 | 294
  Change at Week 2: General Activity | -1.30 (2.58) | -1.72 (2.51) | -2.20 (2.75) | -2.06 (3.00) | -1.92 (2.72)
  Change at Week 4: General Activity: number analyzed (Participants) | 228 | 231 | 295 | 295 | 294
  Change at Week 4: General Activity | -1.33 (2.55) | -2.17 (2.42) | -2.64 (2.59) | -2.90 (2.84) | -2.08 (2.72)
  Change at Week 8: General Activity: number analyzed (Participants) | 228 | 231 | 295 | 295 | 294
  Change at Week 8: General Activity | -1.36 (2.57) | -1.70 (2.52) | -2.27 (2.63) | -2.53 (2.76) | -1.77 (2.64)
  Change at Week 12: General Activity: number analyzed (Participants) | 228 | 231 | 295 | 295 | 294
  Change at Week 12: General Activity | -1.43 (2.54) | -1.76 (2.54) | -2.39 (2.73) | -2.62 (2.87) | -1.90 (2.68)
  Change at Week 16: General Activity: number analyzed (Participants) | 228 | 231 | 295 | 295 | 294
  Change at Week 16: General Activity | -1.34 (2.21) | -1.68 (2.55) | -2.20 (2.76) | -2.26 (2.71) | -1.65 (2.56)
  Change at Week 2: Walking Ability | -1.29 (2.71) | -1.59 (2.52) | -1.83 (2.69) | -1.81 (2.94) | -1.73 (2.71)
  Change at Week 4: Walking Ability | -1.48 (2.71) | -1.91 (2.59) | -2.32 (2.59) | -2.58 (2.88) | -2.00 (2.63)
  Change at Week 8: Walking Ability | -1.24 (2.56) | -1.62 (2.47) | -2.01 (2.66) | -2.36 (2.88) | -1.72 (2.52)
  Change at Week 12: Walking Ability | -1.28 (2.41) | -1.63 (2.50) | -2.13 (2.68) | -2.34 (2.82) | -1.80 (2.55)
  Change at Week 16: Walking Ability | -1.17 (2.16) | -1.49 (2.29) | -1.91 (2.71) | -2.14 (2.72) | -1.53 (2.52)
  Change at Week 2: Normal Work: number analyzed (Participants) | 227 | 231 | 295 | 295 | 294
  Change at Week 2: Normal Work | -1.33 (2.37) | -1.75 (2.57) | -2.01 (2.61) | -2.01 (2.90) | -1.67 (2.67)
  Change at Week 4: Normal Work: number analyzed (Participants) | 227 | 231 | 295 | 295 | 294
  Change at Week 4: Normal Work | -1.59 (2.36) | -2.03 (2.49) | -2.49 (2.57) | -2.79 (2.75) | -2.03 (2.55)
  Change at Week 8: Normal Work: number analyzed (Participants) | 227 | 231 | 295 | 295 | 294
  Change at Week 8: Normal Work | -1.31 (2.35) | -1.72 (2.46) | -2.25 (2.64) | -2.58 (2.75) | -1.76 (2.49)
  Change at Week 12: Normal Work: number analyzed (Participants) | 227 | 231 | 295 | 295 | 294
  Change at Week 12: Normal Work | -1.43 (2.25) | -1.76 (2.43) | -2.35 (2.75) | -2.57 (2.85) | -1.85 (2.65)
  Change at Week 16: Normal Work: number analyzed (Participants) | 227 | 231 | 295 | 295 | 294
  Change at Week 16: Normal Work | -1.27 (2.15) | -1.55 (2.45) | -2.09 (2.74) | -2.40 (2.76) | -1.65 (2.47)
  Change at Week 2: Pain Interference with Sleep | -1.4 (2.72) | -1.7 (2.58) | -2.0 (2.89) | -1.7 (3.09) | -2.2 (2.90)
  Change at Week 4: Pain Interference with Sleep | -1.6 (2.52) | -2.3 (2.62) | -2.6 (2.87) | -2.7 (2.89) | -2.2 (2.72)
  Change at Week 8: Pain Interference with Sleep | -1.4 (2.54) | -1.9 (2.62) | -2.4 (2.86) | -2.4 (2.83) | -1.9 (2.54)
  Change at Week 12: Pain Interference with Sleep | -1.5 (2.49) | -1.8 (2.69) | -2.4 (3.04) | -2.5 (3.00) | -2.0 (2.66)
  Change at Week 16: Pain Interference with Sleep | -1.4 (2.29) | -1.7 (2.66) | -2.3 (3.04) | -2.3 (2.82) | -1.8 (2.60)

9. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
days | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events.

10. Secondary Outcome: Number of Participants With Chronic Low Back Pain (CLBP) Responder Index: Baseline Observation Carried Forward (BOCF)
Description: Chronic Low Back Pain (CLBP) Responder Index: A response was defined as reduction of at least 30% in mean daily average LBPI from baseline to a specified week, decrease of at least 30% in PGA of low back pain from baseline to the specified week and no worsening (increase) in RMDQ total score from baseline to the specified week. Participants who were responders were reported.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
participants
  Week 2 | 38 | 48 | 77 | 80 | 69
  Week 4 | 52 | 70 | 114 | 113 | 79
  Week 8 | 40 | 62 | 96 | 103 | 64
  Week 12 | 45 | 60 | 104 | 105 | 83
  Week 16 | 44 | 52 | 90 | 89 | 63

11. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) at Week 8 and 16
Description: WPAI:SHP is a self-administered questionnaire that measures the effect of general health and symptom severity on work productivity and regular activities. Four scores are derived as percent: activity impairment (AI), impairment while working (IW), overall work impairment (OWI), work time missed (WTM). Each of 4 scores expressed as impairment percentages with a total possible score range of 0 to 100, high percentage= more impairment, less productivity.
Time Frame: Baseline, Week 8, 16
Population: ITT analysis set. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 229 | 232 | 295 | 295 | 295
percentage of impairment
  Baseline: Activity Impairment: number analyzed (Participants) | 228 | 229 | 293 | 295 | 293
  Baseline: Activity Impairment | 58.77 (22.88) | 55.15 (22.63) | 59.32 (21.48) | 60.81 (20.74) | 59.97 (21.27)
  Baseline: Impairment While Working: number analyzed (Participants) | 123 | 120 | 142 | 158 | 145
  Baseline: Impairment While Working | 49.19 (24.85) | 45.17 (23.51) | 49.15 (22.11) | 49.62 (26.01) | 48.90 (24.16)
  Baseline: Overall Work Impairment | 6.29 (21.06) | 6.68 (21.61) | 7.51 (21.18) | 10.71 (26.29) | 8.30 (23.43)
  Baseline: Work Time Missed | 1.97 (8.69) | 3.17 (12.03) | 2.02 (7.22) | 3.82 (11.50) | 3.26 (11.79)
  Change at Week 8: Activity Impairment: number analyzed (Participants) | 190 | 188 | 244 | 236 | 251
  Change at Week 8: Activity Impairment | -14.58 (24.31) | -15.80 (25.16) | -24.96 (26.32) | -27.08 (28.65) | -18.53 (24.08)
  Change at Week 8: Impairment While Working: number analyzed (Participants) | 94 | 93 | 106 | 114 | 112
  Change at Week 8: Impairment While Working | -14.79 (24.79) | -10.75 (25.42) | -21.98 (25.54) | -19.21 (45.39) | -16.70 (23.23)
  Change at Week 8: Overall Work Impairment: number analyzed (Participants) | 193 | 195 | 245 | 241 | 253
  Change at Week 8: Overall Work Impairment | 0.43 (21.56) | 0.08 (19.74) | -3.83 (22.24) | -6.64 (24.52) | -4.58 (20.24)
  Change at Week 8: Work Time Missed: number analyzed (Participants) | 193 | 195 | 245 | 241 | 253
  Change at Week 8: Work Time Missed | 0.58 (8.78) | 0.16 (9.53) | -0.38 (9.12) | -2.15 (12.35) | -1.74 (9.25)
  Change at Week 16: Activity Impairment: number analyzed (Participants) | 128 | 146 | 188 | 190 | 187
  Change at Week 16: Activity Impairment | -22.50 (24.11) | -19.45 (25.51) | -29.95 (27.08) | -31.79 (25.78) | -24.28 (24.62)
  Change at Week 16: Impairment While Working: number analyzed (Participants) | 67 | 69 | 85 | 94 | 86
  Change at Week 16: Impairment While Working | -20.60 (22.56) | -15.22 (24.05) | -27.65 (26.17) | -24.57 (26.34) | -21.05 (24.54)
  Change at Week 16:Overall Work Impairment: number analyzed (Participants) | 128 | 150 | 194 | 193 | 188
  Change at Week 16:Overall Work Impairment | -2.52 (14.15) | -1.72 (15.37) | -3.92 (24.38) | -7.71 (24.10) | -6.68 (22.62)
  Change at Week 16:Work Time Missed: number analyzed (Participants) | 128 | 150 | 194 | 193 | 188
  Change at Week 16:Work Time Missed | -0.79 (6.67) | -0.09 (7.49) | -0.24 (11.20) | -2.98 (10.69) | -2.30 (11.60)

12. Secondary Outcome: Percentage of Participants Who Used Rescue Medications
Description: In case of inadequate pain relief for CLBP or for non-CLBP related pain, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication.
Time Frame: Week 2, 4, 8, 12, 16
Population: ITT analysis set. LOCF method was used to impute missing values. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 293 | 292 | 294
percentage of participants
  Week 2: number analyzed (Participants) | 229 | 231 | 293 | 290 | 291
  Week 2 | 70.3 | 69.7 | 74.1 | 73.4 | 60.8
  Week 4: number analyzed (Participants) | 230 | 232 | 293 | 292 | 293
  Week 4 | 63.9 | 53.9 | 54.3 | 53.4 | 53.2
  Week 8 | 54.8 | 49.6 | 50.9 | 47.6 | 48.3
  Week 12 | 40.4 | 40.5 | 45.1 | 38.7 | 44.6
  Week 16 | 42.6 | 41.4 | 43.0 | 38.0 | 41.2

13. Secondary Outcome: Duration of Rescue Medication Use
Description: as for outcome 12
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 12
Measure: Median (Full Range); unit: days/week
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 293 | 292 | 294
days/week
  Week 2: number analyzed (Participants) | 229 | 231 | 293 | 290 | 291
  Week 2 | 2.0 [0.0 to 7.0] | 2.0 [0.0 to 7.0] | 2.0 [0.0 to 7.0] | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0]
  Week 4: number analyzed (Participants) | 230 | 232 | 293 | 292 | 293
  Week 4 | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0]
  Week 8 | 1.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 12 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 16 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]

14. Secondary Outcome: Amount of Rescue Medication Taken
Description: as for outcome 12
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg per week
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 293 | 292 | 294
mg per week
  Week 2: number analyzed (Participants) | 229 | 231 | 293 | 290 | 291
  Week 2 | 4168.12 (4708.74) | 4305.19 (5102.74) | 3952.22 (4527.82) | 4306.90 (4880.47) | 3350.52 (4564.20)
  Week 4: number analyzed (Participants) | 230 | 232 | 293 | 292 | 293
  Week 4 | 3547.83 (4860.04) | 3252.16 (5189.48) | 2583.62 (3966.56) | 2688.36 (4314.58) | 2680.89 (4120.78)
  Week 8 | 2910.87 (4483.80) | 2633.62 (4309.14) | 2829.35 (4458.51) | 2558.22 (4232.71) | 2477.89 (4270.55)
  Week 12 | 2619.57 (5350.37) | 2256.47 (4350.69) | 2511.95 (4164.31) | 2351.03 (4297.87) | 2455.78 (4580.69)
  Week 16 | 2523.91 (4493.14) | 2140.09 (4167.33) | 2250.85 (3979.75) | 2369.86 (4417.07) | 2448.98 (4677.93)

15. Secondary Outcome: Change From Baseline Neuropathy Impairment Score (NIS) at Week 8, 16 and 24
Description: NIS is a standardized instrument used to evaluate signs of peripheral neuropathy in participants. NIS is the sum of scores of 37 items, from both the left and right side of following 4 domains: cranial nerves (5 items), muscle weakness (19 items), reflexes (5 items) and sensation (8 items). Each of 24 items related to cranial nerves and muscle weakness, scored from 0 (normal) to 4 (paralysis); higher scores indicated higher abnormality/impairment. Each of 13 items related to reflexes and sensation, scored as 0 (normal), 1 (decreased) and 2 (absent); higher scores indicated lesser reflexes and sensation. For NIS possible overall score (combined of both left and right sides of each domain), ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased/more neuropathic deficits.
Time Frame: Baseline, Week 8, 16, 24
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication. Here 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
units on a scale
  Baseline | 0.97 (2.68) | 1.16 (3.04) | 1.03 (2.79) | 1.31 (4.75) | 1.02 (2.82)
  Change at Week 8: number analyzed (Participants) | 193 | 194 | 244 | 240 | 252
  Change at Week 8 | -0.15 (1.43) | -0.41 (2.79) | -0.09 (1.49) | -0.38 (3.61) | -0.06 (1.14)
  Change at Week 16: number analyzed (Participants) | 128 | 150 | 194 | 192 | 188
  Change at Week 16 | -0.30 (1.67) | -0.27 (1.96) | 0.05 (1.36) | 0.02 (1.63) | -0.18 (1.43)
  Change at Week 24: number analyzed (Participants) | 23 | 20 | 21 | 24 | 29
  Change at Week 24 | -0.74 (3.47) | -0.15 (1.09) | 0.10 (1.04) | -0.46 (1.22) | -0.48 (1.48)

16. Secondary Outcome: Number of Participants Who Developed Anti-Tanezumab Antibodies
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). Same participant may have positive ADA result at more than 1 time point.
Time Frame: Baseline (Day 1), Week 8, 16, 24
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication. Here, "Overall number of participants analyzed" = participants who were evaluable for this outcome measure and 'Number Analyzed' = participants who were evaluable for this outcome measure at given time points for each group, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 226 | 288 | 289
Participants
  Baseline | 0 | 1 | 0
  Week 8: number analyzed (Participants) | 173 | 204 | 209
  Week 8 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 135 | 167 | 170
  Week 16 | 0 | 1 | 1
  Week 24: number analyzed (Participants) | 54 | 81 | 80
  Week 24 | 0 | 1 | 1

17. Secondary Outcome: Plasma Concentration of Tanezumab
Description: Analysis was done by setting concentration values below the lower limit of quantification (LLOQ) to zero.
Time Frame: Baseline (pre-dose and 1 hour [hr] post-dose); Any time point at Week 4 Visit; Week 8 (pre-dose and 1 hr post-dose); Any time point at Week 16 Visit, at Week 24 Visit
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 225 | 288 | 288
nanogram per milliliter
  Baseline: pre-dose | 70.7627 (315.3581) | 60.2354 (383.8924) | 40.9396 (317.3858)
  Baseline: 1 hr post-dose: number analyzed (Participants) | 172 | 238 | 243
  Baseline: 1 hr post-dose | 1944.46 (572.9289) | 4105.46 (1495.906) | 8460.14 (2983.547)
  Week 4: number analyzed (Participants) | 190 | 231 | 230
  Week 4 | 472.248 (238.5394) | 983.377 (346.1361) | 1983.72 (598.7860)
  Week 8: pre-dose: number analyzed (Participants) | 171 | 206 | 208
  Week 8: pre-dose | 240.405 (333.2990) | 442.843 (208.6190) | 1081.69 (997.0692)
  Week 8: 1 hr post-dose: number analyzed (Participants) | 155 | 173 | 184
  Week 8: 1 hr post-dose | 2026.01 (693.5790) | 4637.82 (2630.921) | 9161.84 (4274.392)
  Week 16: number analyzed (Participants) | 137 | 174 | 172
  Week 16 | 239.804 (245.3006) | 531.014 (256.1994) | 1393.40 (1219.270)
  Week 24: number analyzed (Participants) | 56 | 82 | 84
  Week 24 | 276.991 (402.0603) | 636.217 (567.9855) | 1222.17 (1105.125)

18. Secondary Outcome: Total Nerve Growth Factor (NGF) Concentration
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: picogram per mL
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 209 | 216 | 277 | 268 | 266
picogram per mL
  Baseline: pre-dose | 34.65 (11.68) | 44.38 (49.12) | 55.66 (202.0) | 61.79 (220.7) | 35.50 (12.38)
  Baseline: 1 hr post-dose: number analyzed (Participants) | 151 | 166 | 211 | 197 | 205
  Baseline: 1 hr post-dose | 37.90 (11.99) | 96.76 (35.08) | 113.33 (251.5) | 126.50 (192.8) | 40.30 (13.10)
  Week 4: number analyzed (Participants) | 142 | 187 | 228 | 231 | 201
  Week 4 | 92.33 (655.1) | 3217.6 (1134) | 3981.7 (1362) | 4456.7 (1325) | 38.17 (16.11)
  Week 8: pre-dose: number analyzed (Participants) | 127 | 173 | 208 | 212 | 191
  Week 8: pre-dose | 126.66 (707.6) | 2671.7 (1249) | 3624.7 (1398) | 4238.6 (1604) | 41.47 (80.11)
  Week 8: 1 hr post-dose: number analyzed (Participants) | 93 | 164 | 196 | 196 | 129
  Week 8: 1 hr post-dose | 124.71 (750.3) | 2943.5 (1334) | 3950.9 (1479) | 4929.1 (1775) | 69.74 (241.8)
  Week 16: number analyzed (Participants) | 99 | 136 | 170 | 171 | 130
  Week 16 | 41.96 (23.56) | 3263.0 (1539) | 4490.5 (1953) | 5842.2 (2377) | 135.17 (810.2)
  Week 24: number analyzed (Participants) | 64 | 54 | 85 | 83 | 77
  Week 24 | 226.61 (916.4) | 2602.0 (1486) | 3549.5 (1747) | 4420.3 (1776) | 38.77 (15.66)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 24 that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Number analyzed (Participants) | 230 | 232 | 295 | 295 | 295
Participants
  AEs | 120 | 141 | 171 | 190 | 142
  SAEs | 5 | 4 | 3 | 3 | 5

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Naproxen 500 mg
Serious Adverse Events (participants affected / at risk) | 5/230 | 4/232 | 3/295 | 3/295 | 5/295
Other Adverse Events (participants affected / at risk) | 74/230 | 80/232 | 114/295 | 134/295 | 76/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=230) | Tanezumab 5 mg (N=232) | Tanezumab 10 mg (N=295) | Tanezumab 20 mg (N=295) | Naproxen 500 mg (N=295)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=230) | Tanezumab 5 mg (N=232) | Tanezumab 10 mg (N=295) | Tanezumab 20 mg (N=295) | Naproxen 500 mg (N=295)
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 8 | 8 | 4
Nausea (Gastrointestinal disorders) | 2 | 6 | 6 | 12 | 9
Oedema peripheral (General disorders) | 2 | 4 | 7 | 10 | 3
Bronchitis (Infections and infestations) | 6 | 5 | 2 | 4 | 3
Influenza (Infections and infestations) | 5 | 6 | 4 | 3 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4 | 10 | 13 | 9
Sinusitis (Infections and infestations) | 5 | 5 | 7 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 10 | 10 | 10 | 12
Urinary tract infection (Infections and infestations) | 8 | 5 | 6 | 11 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 6 | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 26 | 31 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2 | 7 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 9 | 7 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 7 | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6 | 20 | 19 | 2
Dizziness (Nervous system disorders) | 7 | 5 | 2 | 4 | 4
Dysaesthesia (Nervous system disorders) | 2 | 2 | 3 | 8 | 1
Headache (Nervous system disorders) | 9 | 12 | 7 | 13 | 11
Hyperaesthesia (Nervous system disorders) | 2 | 2 | 7 | 12 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 5 | 9 | 10 | 8
Paraesthesia (Nervous system disorders) | 5 | 11 | 21 | 38 | 5
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 8

LIMITATIONS AND CAVEATS:
Results for total duration of response as defined by days with a >=30% and a >=50% reduction from baseline in the daily average LBPI NRS score was not reported due changed in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.